CLINICAL TRIAL: NCT00519142
Title: A Rapid Onset and Short Duration Insulin Secretogogue, Mitiglinide, in Combination With Metformin Versus Metformin Alone in Patients With Type 2 Diabetes Mellitus: A Randomized, Double-blind, Placebo-controlled Trial for 6 Months
Brief Title: Mitiglinide in Combination With Metformin vs. Metformin Alone in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Elixir Pharmaceuticals (Industry)
Responsible Party: Paul Martha, Chief Medical Officer, Elixir Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EX-1510-CT-003
Record Dates: First submitted 2007-08-20; First posted 2007-08-22 (Estimated); Last update posted 2009-09-17 (Estimated); Status verified 2009-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — mitiglinide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): metformin + placebo for mitiglinide
  Interventions: Drug: placebo for mitiglinide
- 2 (Experimental): metformin + mitiglinide three times a day with meals
  Interventions: Drug: mitiglinide
- 3 (Experimental): metformin + mitiglinide two times a day with morning and evening meal, placebo for mitiglinide with midday meal
  Interventions: Drug: mitiglinide

INTERVENTIONS:
Drug: placebo for mitiglinide — three times a day with meals
  Arms: 1
Drug: mitiglinide — three times a day with meals
  Arms: 2
Drug: mitiglinide — two times a day with meals
  Arms: 3

SUMMARY:
The primary objective of this study is to demonstrate whether mitiglinide administered in combination with metformin is more effective than metformin alone in patients with Type 2 diabetes mellitus (T2DM) whose blood sugar is not well controlled taking metformin alone. This is a 24 week study which measures improvement in blood sugar after of treatment.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel group study designed to evaluate the efficacy and safety of mitiglinide in combination with metformin in patients with T2DM who are less than adequately controlled on metformin alone. Patients who are receiving metformin alone for T2DM will be randomized equally into one of three treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes diagnosed for at least 6 months
* stable metformin usage for at least 4 months
* HbA1c 7.5% - 10.5% inclusive
* no severe diabetic complications

Exclusion Criteria:

* chronic insulin use
* use of oral diabetic agent within 12 weeks
* acute or chronic conditions, excluding diabetes, that could compromise end point evaluation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 367 (Actual)
Dates: Start 2007-08; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
change from baseline in HbA1c | after 24 weeks of treatment

SECONDARY OUTCOMES:
change from baseline in 2-hour post-prandial glucose | after 24 weeks of treatment
change from baseline in fasting plasma glucose | after 24 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Paul Martha, MD, Study Director — Elixir Pharmaceuticals
Locations (61):
- United States (57):
  - Elixir Study Site, Glendale, Arizona
  - Elixir Study Site, Greenbrae, California
  - Elixir Study Site, La Jolla, California
  - Elixir Study Site, Los Angeles, California
  - Elixir Study Site, Los Gatos, California
  - Elixir Study Site(s), Oakland Area, California
  - Elixir Study Site, Orange, California
  - Elixir Study Site, West Hills, California
  - Elixir Study Site, Westlake Village, California
  - Elixir Study Site, Pueblo, Colorado
  - Elixir Study Site(s), Washington D.C., District of Columbia
  - Elixir Study Site, Chiefland, Florida
  - Elixir Study Site, Coral Gables, Florida
  - Elixir Study Site, Kissimmee, Florida
  - Elixir Study Site(s), Miami, Florida
  - Elixir Study Site, Saint Cloud, Florida
  - Elixir Study Site, Winter Park, Florida
  - Elixir Study Site, Atlanta, Georgia
  - Elixir Study Site, Austell, Georgia
  - Elixir Study Site, Perry, Georgia
  - Elixir Study Site(s), Chicago, Illinois
  - Elixir Study Site, Wichita, Kansas
  - Elixir Study Site, Kansas City, Missouri
  - Elixir Study Site, St Louis, Missouri
  - Elixir Study Site, Las Vegas, Nevada
  - Elixir Study Site, Hamilton, New Jersey
  - Elixir Study Site, Hillsborough, New Jersey
  - Elixir Study Site, Sewell, New Jersey
  - Elixir Study Site(s), New York, New York
  - Elixir Study Site, Mooresville, North Carolina
  - Elixir Study Site, Morehead City, North Carolina
  - Elixir Study Site, Akron, Ohio
  - Elixir Study Site, Cincinnati, Ohio
  - Elixir Study Site, Gallipolis, Ohio
  - Elixir Study Site, Kettering, Ohio
  - Elixir Study Site, Medford, Oregon
  - Elixir Study Site, Harleysville, Pennsylvania
  - Elixir Study Site, Levittown, Pennsylvania
  - Elixir Study Site, Uniontown, Pennsylvania
  - Elixir Study Site, Columbia, South Carolina
  - Elixir Study Site, Simpsonville, South Carolina
  - Elixir Study Site, Memphis, Tennessee
  - Elixir Study Site, Tullahoma, Tennessee
  - Elixir Study Site(s), Dallas, Texas
  - Elixir Study Site, El Paso, Texas
  - Elixir Study Site(s), Fort Worth, Texas
  - Elixir Study Site(s), Houston, Texas
  - Elixir Study Site, Humble, Texas
  - Elixir Study Site, Midland, Texas
  - Elixir Study Site, New Braunfels, Texas
  - Elixir Study Site, North Richland Hills, Texas
  - Elixir Study Site, Pearland, Texas
  - Elixir Study Site, Plano, Texas
  - Elixir Study Site(s), San Antonio, Texas
  - Elixir Study Site, Temple, Texas
  - Elixir Study Site, Norfolk, Virginia
  - Elixir Study Site, Federal Way, Washington
- Puerto Rico (4):
  - Elixir Study Site, Carolina
  - Elixir Study Site, Fajardo
  - Elixir Study Site(s), Ponce
  - Elixir Study Site(s), San Juan